CLINICAL TRIAL: NCT02830269
Title: Third Ventricle Echographic Study for Neuro-intensive Care Unit Patients
Acronym: ECHO-V3
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9720; 2016-A00749-42 (Other: RCB number)
Record Dates: First submitted 2016-06-10; First posted 2016-07-12 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2017-04

CONDITIONS: Neuro-intensive Care Unit Patients; Brain Injuries
Keywords: Neuro-ICU; Third ventricle; Computer Tomography; Transcranial Doppler ultrasonography
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Transcranial Doppler ultrasonography measurements — Third ventricle diameter measurements with standard method (CT) and Transcranial Doppler ultrasonography

SUMMARY:
Transcranial Doppler ultrasonography is usually used in the evaluation and management of patients with brain injury. This noninvasive method measures local blood flow velocity and direction in the proximal portions of large intracranial arteries. The operator requires a short training and experience to perform. The third ventricle diameter measurement by transcranial duplex flow sonography was performed in healthy volunteers . This studies show similar results in those obtained with the MRI or Computer Tomography (CT). Currently the third ventricle diameter measurements by transcranial Doppler ultrasonography was not validated for neuro-intensive care unit patients. The investigators propose to used recent ultrasound system to validate the third ventricle diameter measurements in comparison with the standard method (CT).

DETAILED DESCRIPTION:
Transcranial Doppler ultrasonography is usually used in the evaluation and management of patients with brain injury. This noninvasive method measures local blood flow velocity and direction in the proximal portions of large intracranial arteries. The operator requires a short training and experience to perform. The third ventricle diameter measurement by transcranial duplex flow sonography was performed in healthy volunteers . This studies show similar results in those obtained with the MRI or Computer Tomography (CT). Currently the third ventricle diameter measurements by transcranial Doppler

ELIGIBILITY:
Inclusion Criteria:

* Adult, > or equal to 18-yr
* Admission to neuro-intensive care unit with brain injury
* Evaluation by Computer Tomography
* Indication for Transcranial Doppler ultrasonography

Exclusion Criteria:

* Opposition to participate by the patient or a next of kin

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the neurointensive care
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Third ventricle diameter (average +/- standard deviation) | Through study completion (30 months)
  Spearman's test measuring the correlation coefficient between the third ventricle diameter measured by the expert using the ultrasonography and the third ventricle diameter measured by CT scan.

SECONDARY OUTCOMES:
Residents' learning curve | 24 months
  The learning curve will be determined by the change in the third ventricle diameter's difference obtained by the expert and the resident, divided by the diameter obtained by the expert reported on the Y-axis and the number of measures done by the resident reported on the X-axis. Number of measures to be done will be determined when the curve reached the zero.

CONTACTS AND LOCATIONS:
Overall Officials: GERALD CHANQUES, MD, Ph D, Study Director — University Hospital, Montpellier; Pierre-François PERRIGAULT, MD, Study Chair — University Hospital, Montpellier; Paul BORY, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

REFERENCES:
- [Derived] Widehem R, Bory P, Greco F, Pavillard F, Chalard K, Mas A, Djanikian F, Carr J, Molinari N, Jaber S, Perrigault PF, Chanques G. Transcranial sonographic assessment of the third ventricle in neuro-ICU patients to detect hydrocephalus: a diagnostic reliability pilot study. Ann Intensive Care. 2021 May 4;11(1):69. doi: 10.1186/s13613-021-00857-x. PMID 33945045